CLINICAL TRIAL: NCT00815516
Title: A Phase 3, Randomized, Double-Blind, Multi-Center Study to Compare the Efficacy and Safety of Micafungin Versus Amphotericin B Deoxycholate for the Treatment of Neonatal Candidiasis
Brief Title: Study to Compare the Efficacy and Safety of Micafungin Versus Conventional Amphotericin B for the Treatment of Neonatal Candidiasis
Acronym: MAGIC-2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: It was decided to discontinue the study due to insufficient recruitment.
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9463-CL-2303; 2012-000780-24 (EudraCT Number)
Record Dates: First submitted 2008-12-27; First posted 2008-12-30 (Estimated); Results first posted 2015-09-15 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-10

CONDITIONS: Candidiasis
Keywords: candidiasis; candida; Neonate; candidemia; Micafungin; Mycamine; amphotericin B deoxycholate
MeSH Terms: conditions — Candidiasis; Torulopsis; Candidemia | interventions — Micafungin; amphotericin B, deoxycholate drug combination; Amphotericin B; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Micafungin (Experimental): Infants received micafungin at a dose of 10 mg/kg per day by intravenous infusion for a minimum of 21 days to a maximum of 28 days for infants without end-organ dissemination or for a maximum of 42 days for infants with end-organ dissemination.
  Interventions: Drug: micafungin
- Amphotericin B deoxycholate (Active Comparator): Infants received amphotericin B deoxycholate (CAB) at a dose of 1.0 mg/kg per day by intravenous infusion for a minimum of 21 days to a maximum of 28 days for infants without end-organ dissemination or for a maximum of 42 days for infants with end-organ dissemination.
  Interventions: Drug: amphotericin B deoxycholate

INTERVENTIONS:
Drug: micafungin — Administered by intravenous infusion
  Other Names: Mycamine; FK463
  Arms: Micafungin
Drug: amphotericin B deoxycholate — Administered by intravenous infusion
  Other Names: Fungizone; Conventional amphotericin B (CAB); Amphotericin B for injection
  Arms: Amphotericin B deoxycholate

SUMMARY:
The study will evaluate how effective and how safe the drug micafungin is when compared to the drug amphotericin B deoxycholate in treating neonates and young infants with certain fungal infections.

DETAILED DESCRIPTION:
Neonates and young infants will be stratified by estimated gestational age and by world region

ELIGIBILITY:
Inclusion Criteria:

* Infant greater than 48 hours of life after birth up to day of life 120 at the time of culture acquisition
* Diagnosis of proven invasive candidiasis within 4 days prior to study start
* Subject's parent or legal guardian agrees not to allow subject to participate in another study with another investigational drug while on treatment.

Exclusion Criteria:

* Infant with any history of a hypersensitivity or severe vasomotor reaction to any echinocandin or systemic amphotericin B product
* Infant who has received more than 48 hours of systemic antifungal therapy prior to the first dose of study drug
* Infant who has a breakthrough systemic fungal infection while receiving amphotericin B product or an echinocandin as prophylaxis
* Infant who has failed prior systemic antifungal therapy for this episode of invasive candidiasis
* Infant who is co-infected with a non-Candida fungal organism
* Infant whose positive yeast cultures are solely from an indwelling bladder catheter (unless obtained at the time the indwelling catheter was placed) or sputum.
* Infant previously enrolled in this study

Ages: 48 Hours to 120 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2013-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development
Locations (17):
- United States (5):
  - Children's Hospital of Orange County, Orange, California
  - UMDNJ/Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Duke University, Durham, North Carolina
  - WakeMed Health and Hospitals, Raleigh, North Carolina
  - Virginia Commonwealth University, Richmond, Virginia
- Brazil (2):
  - Irmandade da Santa Casa de Misericórdia de Belo Horizonte, Belo Horizonte, Minas Gerais
  - Hospital de Base da Faculdade de Medicina, São José do Rio Preto, São Paulo
- Spec Hospital for Active Treatment of Children Diseases, Sofia, Bulgaria
- McMaster Children's Hospital, Hamilton, Ontario, Canada
- Hospital Pablo Tobon Uribe, Medellín, Antioque, Colombia
- University Hospital of Patras, Pátrai, Greece
- Semmelweis Egyetem, Budapest, Hungary
- Hadassah University Hospital Ein Kerem, Jerusalem, Israel
- Philippine General Hospital, Manila, Philippines
- Emergency County Clinical Hospital, Cluj-Napoca, Romania
- Cukurova University Medical Faculty, Adana, Turkey (Türkiye)
- Municipal Institution "Odesa Regional Children's Hospital", Odesa, Ukraine

REFERENCES:
- [Derived] Benjamin DK Jr, Kaufman DA, Hope WW, Smith PB, Arrieta A, Manzoni P, Kovanda LL, Lademacher C, Isaacson B, Jednachowski D, Wu C, Kaibara A, Walsh TJ. A Phase 3 Study of Micafungin Versus Amphotericin B Deoxycholate in Infants With Invasive Candidiasis. Pediatr Infect Dis J. 2018 Oct;37(10):992-998. doi: 10.1097/INF.0000000000001996. PMID 29596222
- See also: Link to results on Astellas Clinical Study Results Web site — https://www.astellasclinicalstudyresults.com/study.aspx?ID=9463-CL-2303

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Infants greater than 48 hours of life through day of life (DOL) 120 with a diagnosis of invasive candidiasis were eligible for this study.
Pre-assignment Details: In total, 31 infants were screened and 30 were randomized in a 2:1 ratio to receive micafungin or amphotericin B deoxycholate. Randomization was stratified by estimated gestational age (< 27 weeks, ≥ 27 weeks) and by region (North America/Europe, Latin America / Mexico, other region).
Groups:
- Amphotericin B: Infants received amphotericin B deoxycholate (CAB) at a dose of 1.0 mg/kg per day by intravenous infusion for a minimum of 21 days to a maximum of 28 days for infants without end-organ dissemination or for a maximum of 42 days for infants with end-organ dissemination.
Period: Overall Study
Arm/Group | Micafungin | Amphotericin B
Started | 20 | 10
Completed | 16 | 9
Not Completed | 4 | 1
Not completed — Death | 3 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Micafungin | Amphotericin B | Total
Number analyzed (Participants) | 20 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: days] | 30.2 (27.99) | 16.9 (5.13) | 25.7 (23.70)
Age, Customized [Number; unit: participants]
  ≤ 4 weeks | 15 | 10 | 25
  > 4 weeks to 4 months | 5 | 0 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 4 | 16
  Male | 8 | 6 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 4 | 3 | 7
  Unknown or Not Reported | 13 | 4 | 17
Race/Ethnicity, Customized [Number; unit: participants]
  White | 18 | 9 | 27
  Black or African American | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Other | 1 | 0 | 1
Gestational Age [Number; unit: participants]
  < 27 Weeks | 3 | 2 | 5
  ≥ 27 Weeks | 17 | 8 | 25
Region of Enrollment [Number; unit: participants]
  North America /Europe | 15 | 9 | 24
  Latin America /Mexico | 4 | 1 | 5
  Other | 1 | 0 | 1
Birth Weight [Mean (Standard Deviation); unit: grams] | 1807.3 (879.03) | 2171.4 (1008.79) | 1928.6 (923.34)
Fungal Infection Type [Number; unit: participants] — Candidemia: diagnosed if Candida isolated from blood only; Invasive candidiasis: diagnosed if Candida isolated from blood in addition to other body fluids such as cerebrospinal fluid (CSF), peritoneal fluid, or urine.
  participants
    Candidemia | 12 | 7 | 19
    Invasive Candidiasis | 8 | 2 | 10
    Missing | 0 | 1 | 1
Presence of End-Organ Dissemination (EOD) [Number; unit: participants] — End-organ dissemination was assessed using echocardiogram, abdominal ultrasound, including evaluation of the liver, spleen, and kidneys, head ultrasound, computed tomography (CT) or magnetic resonance imaging (MRI), and retinal exam (if clinically feasible). End-organ dissemination was assessed by the data review panel (DRP). Missing for the DRP assessment means that no evidence for EOD was documented.
  participants
    Yes | 7 | 3 | 10
    Missing | 13 | 7 | 20

OUTCOME MEASURES:

1. Primary Outcome: Fungal-free Survival
Description: Fungal-free survival was assessed by an independent data review panel (DRP). Fungal-free survival is defined as the percentage of participants alive at one week following the last dose of study drug with a mycological response of eradication and no requirement for alternative systemic antifungal therapy for continued treatment.
  Eradication was defined as culture or histologically documented absence of the infecting Candida species from all positive normally sterile sites during therapy, documented by 2 negative samples, drawn at least 24 hours apart, or for Candida meningitis and/or candiduria, 1 negative culture.
Time Frame: One week after the last dose of study drug (maximum of 49 days)
Population: Full Analysis Set (all randomized infants who were administered any amount of study drug)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Micafungin | Amphotericin B
Number analyzed (Participants) | 20 | 10
percentage of participants | 60.0 [36.1 to 80.9] | 70.0 [34.8 to 93.3]

2. Secondary Outcome: Time to Mycological Clearance of Invasive Candidiasis
Description: Time to mycological clearance of invasive candidiasis is defined as the time from first dose to the day of mycological eradication for baseline invasive candidiasis infection.
  Eradication was defined as a culture or histologically documented absence of the infecting Candida species from all positive normally sterile sites during therapy, documented by 2 negative samples, drawn at least 24 hours apart, or for for Candida meningitis and/or candiduria, 1 negative culture.
  Infants without eradication during the treatment period and who survived were censored at one day after the end of treatment. Infants without eradication who died before completing the treatment period or were lost to follow-up during the treatment were censored at their death or last contact day.
Time Frame: From first dose up to 30 days after the last dose of study drug (maximum of 72 days)
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Micafungin | Amphotericin B
Number analyzed (Participants) | 20 | 10
days | 6.0 [3.0 to NA] — Could not be estimated due to the low number of events. | 3.0 [0.0 to 9.0]

3. Secondary Outcome: Fungal-free Survival at End of Study Drug Therapy in Infants With End-organ Dissemination
Description: Fungal-free survival was assessed by an independent data review panel (DRP). Fungal-free survival is defined as the percentage of participants alive at the end of study drug therapy with a mycological response of eradication based upon the DRP assessment and no requirement for alternative systemic antifungal therapy for continued treatment.
Time Frame: The end of study drug therapy; maximum of 42 days
Population: Participants in the full analysis set with end-organ dissemination
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Micafungin | Amphotericin B
Number analyzed (Participants) | 7 | 3
percentage of participants | 42.9 [9.9 to 81.6] | 33.3 [0.8 to 90.6]

4. Secondary Outcome: Fungal-free Survival One Week After Last Dose of Study Drug in Infants With End-organ Dissemination
Description: Fungal-free survival was assessed by an independent data review panel (DRP). Fungal-free survival is defined as the percentage of participants alive one week after last dose of study drug with a mycological response of eradication based upon the DRP assessment and no requirement for alternative systemic antifungal therapy for continued treatment.
Time Frame: One week after the last dose of study drug (maximum of 49 days)
Population: Participants in the full analysis set with end-organ dissemination
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Micafungin | Amphotericin B
Number analyzed (Participants) | 7 | 3
percentage of participants | 42.9 [9.9 to 81.6] | 33.3 [0.8 to 90.6]

5. Secondary Outcome: Percentage of Participants With Emergent Fungal Infections
Description: An emergent fungal infection is defined as
  * An invasive fungal infection which is detected at any time during the study that is a non-Candida organism, or
  * An invasive fungal infection which is detected during the treatment or post-treatment period with a Candida species identified other than those detected at Baseline. If this occurred within 96 hours of the first dose of study drug, the infection was considered part of the final diagnosis of enrolling infection and not an emergent infection.
Time Frame: Up to 30 days after the last dose of study drug (maximum of 72 days)
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Micafungin | Amphotericin B
Number analyzed (Participants) | 20 | 10
percentage of participants | 5.0 [0.1 to 24.9] | 0 [NA to NA] — Could not be calculated since there were no events in this group

6. Secondary Outcome: Percentage of Participants With Recurrent Fungal Infections
Description: A recurrent infection is defined as a systemic fungal infection in an infant with eradication at the end of study drug therapy, who developed positive blood cultures or a mycologically confirmed deep-seated Candida infection, with the same species as the enrolling infection.
Time Frame: Up to 30 days after the last dose of study drug (maximum of 72 days)
Population: Participants in the full analysis set with eradication at the end of study drug therapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Micafungin | Amphotericin B
Number analyzed (Participants) | 11 | 8
percentage of participants | 0 [NA to NA] — Could not be calculated since there were no events in this group | 12.5 [0.3 to 52.7]

7. Secondary Outcome: Time to Positive Clinical Response
Description: Time to a positive clinical response is defined as the time from the first dose to the day during the treatment period that a positive clinical response (defined as a complete response or partial response) is observed for the first time, assessed by the Investigator.
  Complete Response is defined as the resolution of all attributable signs related to fungal infection, if present at baseline and Partial Response is defined as improvement in attributable signs related to the fungal infection, if present at baseline.
  Infants without positive responses and who survived were censored at one day post the end of treatment. Infants without positive responses who died before completing the treatment period, or were lost to follow-up during the treatment were censored at their death or last contact day.
Time Frame: From first dose up to 30 days after the last dose of study drug (maximum of 72 days)
Population: Full analysis set participants with clinical signs and symptoms related to the fungal Infection at Baseline
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Micafungin | Amphotericin B
Number analyzed (Participants) | 18 | 10
days | 8.0 [7.0 to 15.0] | 11.0 [7.0 to 14.0]

8. Secondary Outcome: Clinical Response at the End of Study Drug Therapy
Description: Clinical response assessments were based on the following definitions and assessed by the DRP:
  * Complete Response: Resolution of all attributable signs related to fungal infection, if present at baseline.
  * Partial Response: Improvement in attributable signs related to the fungal infection, if present at baseline.
  * Stabilization: Minor improvement or no change in attributable signs related to the fungal infection, if present at baseline, and infant continued on therapy without deterioration.
  * Progression: Deterioration in attributable signs related to the fungal infection, if present at baseline; or if death occurred presumably related to a fungal infection.
Time Frame: Baseline and end of study drug therapy; maximum of 42 days
Population: Full analysis set participants with clinical signs and symptoms related to the fungal Infection at Baseline
Measure: Number; unit: percentage of participants
Arm/Group | Micafungin | Amphotericin B
Number analyzed (Participants) | 18 | 10
percentage of participants
  Complete | 55.6 | 70.0
  Partial | 5.6 | 0
  Stable | 5.6 | 10.0
  Progression | 16.7 | 20.0
  Missing | 16.7 | 0

9. Secondary Outcome: Clinical Response One Week After Last Dose of Study Drug
Description: as for outcome 8
Time Frame: Baseline and one week after the last dose of study drug (maximum of 49 days)
Population: Full analysis set participants with clinical signs and symptoms related to the fungal Infection at Baseline
Measure: Number; unit: percentage of participants
Arm/Group | Micafungin | Amphotericin B
Number analyzed (Participants) | 18 | 10
percentage of participants
  Complete | 55.6 | 70.0
  Partial | 5.6 | 0
  Stable | 5.6 | 10.0
  Progression | 5.6 | 20.0
  Missing | 27.8 | 0

10. Secondary Outcome: Mycological Response at End of Study Drug Therapy
Description: Mycological response assessments were based on the following definitions and assessed by the DRP:
  * Eradication: Culture or histologically documented absence of the infecting Candida species from all positive normally sterile sites during therapy, documented by 2 negative samples, drawn at least 24 h apart; for Candida meningitis and/or candiduria, 1 negative culture.
  * Persistence: Continued isolation or histological documentation from a normally sterile site.
Time Frame: End of study drug therapy; maximum of 42 days
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Micafungin | Amphotericin B
Number analyzed (Participants) | 20 | 10
percentage of participants
  Eradication | 55.0 | 80.0
  Persistence | 10.0 | 20.0
  Not Assessed | 35.0 | 0

11. Secondary Outcome: Mycological Response One Week After Last Dose of Study Drug
Description: as for outcome 10
Time Frame: One week after the last dose of study drug (maximum of 49 days)
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Micafungin | Amphotericin B
Number analyzed (Participants) | 20 | 10
percentage of participants
  Continuing Eradication/Eradication | 55.0 | 80.0
  Persistence | 10.0 | 20.0
  Not Assessed | 35.0 | 0

12. Secondary Outcome: Follow-up Status for Infants With End-organ Assessments
Description: End-organ dissemination was assessed through abdominal ultrasound and/or computed tomography (CT), echocardiogram, head imaging and retinal exam. Each specific finding, documented by 1 of these techniques, was evaluated as follows:
  * Improvement: Improvement in size, number or density of identified lesions. Complete response was not expected but may have been documented.
  * Stabilization: Minor improvement or no change in size, number or density of identified lesions.
  * Worsening: Increase in size or number of identified lesions.
Time Frame: Baseline and 30 days after the last dose of study drug (maximum of 72 days)
Population: Full analysis set participants with end-organ assessments
Measure: Number; unit: percentage of participants
Arm/Group | Micafungin | Amphotericin B
Number analyzed (Participants) | 7 | 3
percentage of participants
  Improved | 57.1 | 33.3
  Stable | 14.3 | 0
  Worsened | 14.3 | 66.7
  Not Assessed | 14.3 | 0

13. Secondary Outcome: Plasma Micafungin Concentration
Time Frame: 15 minutes post intravenous infusion (IV), 4-8 hours post IV and 15-24 hours post IV
Population: The pharmacokinetics (PK) analysis set, including those infants who received any amount of study drug, have at least one study drug concentration, and have dosing and blood collection date and time data sufficient for inclusion in a population pharmacokinetic analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Micafungin
Number analyzed (Participants) | 12
ng/mL
  Within 15 Minutes Post IV | 25130.5 (13964.3)
  4-8 Hours Post IV | 23751.7 (9547.7)
  15-24 Hours Post IV | 14118.3 (12396.0)

ADVERSE EVENTS:
Time Frame: From first dose of study drug until 72 hours after the last dose; mean duration of study drug exposure among micafungin-treated patients was 18.6 days and 15.5 days for Amphotericin B-treated patients.
Arm/Group | Micafungin | Amphotericin B
Serious Adverse Events (participants affected / at risk) | 12/20 | 7/10
Other Adverse Events (participants affected / at risk) | 14/20 | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Micafungin (N=20) | Amphotericin B (N=10)
Sepsis (Infections and infestations) | 1 | 1
Sepsis neonatal (Infections and infestations) | 0 | 2
Septic shock (Infections and infestations) | 2 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 4 | 1
Cardiovascular insufficiency (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Oliguria (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Hypothermia (General disorders) | 0 | 1
Hydrocephalus (Nervous system disorders) | 1 | 0
Intraventricular haemorrhage (Nervous system disorders) | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Micafungin (N=20) | Amphotericin B (N=10)
Anaemia (Blood and lymphatic system disorders) | 5 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 3
Neutropenia (Blood and lymphatic system disorders) | 3 | 0
Anaemia neonatal (Blood and lymphatic system disorders) | 1 | 1
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Staphylococcal infection (Infections and infestations) | 2 | 0
Urinary tract infection bacterial (Infections and infestations) | 2 | 0
Endocarditis (Infections and infestations) | 1 | 0
Neonatal infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Pyrexia (General disorders) | 1 | 2
Hypothermia (General disorders) | 1 | 0
Infusion related reaction (General disorders) | 0 | 1
Infusion site extravasation (General disorders) | 0 | 1
Infusion site rash (General disorders) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Antithrombin III decreased (Investigations) | 0 | 1
Bacteria blood identified (Investigations) | 1 | 0
Blood bilirubin abnormal (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Blood urea increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Hepatic enzyme abnormal (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0
Neutrophil count increased (Investigations) | 0 | 1
Oxygen consumption increased (Investigations) | 0 | 1
Serum ferritin increased (Investigations) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Medical device complication (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1
Intraventricular haemorrhage (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1
Galactorrhoea (Reproductive system and breast disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data or 18 months after data-lock, whichever is first. Sponsor must receive a site's manuscript at least 30 days prior to publication for review and comment. Sponsor may delay the publication for up to 60 days to seek patent protection.